CLINICAL TRIAL: NCT01340781
Title: Evaluation of Screening Tools for OSA in Hospitalized Medical Patients: A Validation Study
Brief Title: Screening Tools for Obstructive Sleep Apnea (OSA) in Hospitalized Medical Patients
Acronym: STOMP
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Dennis Auckley, MD, Director, Center for Sleep Medicine, MetroHealth Medical Center
Other Study IDs: Cephalon-01736
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: inpatients; medical; polysomnogram; questionnaires
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hospitalized medical patients: Adult age 18-65 years old admitted to the general medical floors at MetroHealth Medical Center who are expected to stay a minimum of 48 hours.
  Potential subjects cannot have a known diagnosis of OSA, a tracheostomy, respiratory failure requiring noninvasive ventilation, currently pre or post surgical intervention, or clinically unstable patients with plans for transfer to a higher acuity of care or transferred from intensive care.
  Interventions: Procedure: Polysomnogram

INTERVENTIONS:
Procedure: Polysomnogram — An attended polysomnogram will be conducted in the subjects room during an in patient hospital stay

SUMMARY:
The prevalence of obstructive sleep apnea (OSA) in patients admitted to the hospital is likely significantly higher than the general population as hospitalized patients carry a high prevalence of co-morbid conditions, such as diabetes and cardiovascular diseases, that are commonly associated with OSA. The true prevalence of OSA in hospitalized patients is not known, though there is limited data suggesting that the rate of OSA in hospitalized patients is indeed high. Two studies have reported on the rate of polysomnographic (PSG) diagnosis of OSA in patients referred for OSA evaluation while in-hospital. These studies reported frequencies of 77% (in a retrospective study of 100 patients) and 88-100% (in an observational study of 250 patients). Similarly, 2 studies evaluated the prevalence of sleep disordered breathing in patients admitted with acutely decompensated heart failure, finding frequencies of sleep apnea in 97% (prospective study of 29 patients studied with PSG) and 75% (prospective study of 395 consecutive patients studied with portable monitors). However, all of these studies are limited by either study design (retrospective), small numbers, limited channel portable monitoring, or evaluations of highly select patient populations. Furthermore, none of these studies examined screening tools that may help to identify which patients are at risk for OSA and thus might require the more extensive and expensive objective testing.

This study will test the following hypotheses:

1. The prevalence of OSA in unselected hospitalized medical patients will be more than 50% of the study population.

   Specific Aim 1: To determine the prevalence of OSA in a group of unselected hospitalized medical patients by a combination of sleep symptoms and PSG performed while in-hospital.
2. Screening tools will be able to accurately identify OSA in hospitalized medical patients.

Specific Aim 2: To determine the accuracy of different screening questionnaires for the diagnosis of OSA in hospitalized medical patients by comparing the questionnaire results to that of a PSG performed while in-hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-65 years old
* Admitted to the general medical floors at MetroHealth Medical Center
* Expected stay of 48 hours
* Competent to sign informed consent
* Agreeable to participating in the study

Exclusion Criteria:

* Known OSA
* Patients with a tracheostomy
* Clinically unstable patients with plans for transfer to a higher acuity of care
* Patients with planned surgical interventions or status post operation during the admission
* Patients transferred from intensive care
* Patients with respiratory failure requiring noninvasive ventilation
* Inability to comprehend or complete the questionnaires
* Inability to tolerate a sleep study (i.e. allergic to testing components, refusal to wear leads)
* Refusal to sign consent
* Non-English speaking patients
* In an isolation room

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized medical patients
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of OSA in a group of unselected hospitalized medical patients by a combination of sleep symptoms and PSG performed while in-hospital. | 1 year
  Subjects will complete an overnight polysomnogram during an inpatient admission. Data from the PSG will be used to determine if the subject has sleep apnea.

SECONDARY OUTCOMES:
To determine the accuracy of different screening questionnaires for the diagnosis of OSA in hospitalized medical patients by comparing the questionnaire results to that of a PSG performed while in-hospital. | 1 year
  Subjects will complete 4 questionnaires (Berlin, STOP, STOP-BANG, SACS) used to assess risk for OSA prior to polysomnogram testing. The PSG data will be compared to the questionnaire results to determine the validity of the screening questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis H Auckley, M.D., Principal Investigator — MetroHealth System, Ohio
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Hiestand DM, Britz P, Goldman M, Phillips B. Prevalence of symptoms and risk of sleep apnea in the US population: Results from the national sleep foundation sleep in America 2005 poll. Chest. 2006 Sep;130(3):780-6. doi: 10.1378/chest.130.3.780. PMID 16963675
- [Background] Goring K, Collop N. Sleep disordered breathing in hospitalized patients. J Clin Sleep Med. 2008 Apr 15;4(2):105-10. PMID 18468307
- [Background] Al-Jawder S, Bahammam A. Utility of daytime polysomnography for in-patients with suspected sleep-disordered breathing. Neurol Neurochir Pol. 2009 Mar-Apr;43(2):140-7. PMID 19484691
- [Background] Padeletti M, Green P, Mooney AM, Basner RC, Mancini DM. Sleep disordered breathing in patients with acutely decompensated heart failure. Sleep Med. 2009 Mar;10(3):353-60. doi: 10.1016/j.sleep.2008.03.010. Epub 2008 Jul 9. PMID 18614398
- [Background] Khayat RN, Jarjoura D, Patt B, Yamokoski T, Abraham WT. In-hospital testing for sleep-disordered breathing in hospitalized patients with decompensated heart failure: report of prevalence and patient characteristics. J Card Fail. 2009 Nov;15(9):739-46. doi: 10.1016/j.cardfail.2009.05.005. Epub 2009 Jun 26. PMID 19879459
- [Background] Spurr KF, Graven MA, Gilbert RW. Prevalence of unspecified sleep apnea and the use of continuous positive airway pressure in hospitalized patients, 2004 National Hospital Discharge Survey. Sleep Breath. 2008 Aug;12(3):229-34. doi: 10.1007/s11325-007-0166-2. Epub 2008 Jan 31. PMID 18236092
- [Background] Namen AM, Wymer A, Case D, Haponik EF. Performance of sleep histories in an ambulatory medicine clinic: impact of simple chart reminders. Chest. 1999 Dec;116(6):1558-63. doi: 10.1378/chest.116.6.1558. PMID 10593776
- [Background] Haponik EF, Frye AW, Richards B, Wymer A, Hinds A, Pearce K, McCall V, Konen J. Sleep history is neglected diagnostic information. Challenges for primary care physicians. J Gen Intern Med. 1996 Dec;11(12):759-61. doi: 10.1007/BF02598994. PMID 9016425
- [Background] Reuveni H, Tarasiuk A, Wainstock T, Ziv A, Elhayany A, Tal A. Awareness level of obstructive sleep apnea syndrome during routine unstructured interviews of a standardized patient by primary care physicians. Sleep. 2004 Dec 15;27(8):1518-25. doi: 10.1093/sleep/27.8.1518. PMID 15683143
- [Background] Namen AM, Landry SH, Case LD, McCall WV, Dunagan DP, Haponik EF. Sleep histories are seldom documented on a general medical service. South Med J. 2001 Sep;94(9):874-9. PMID 11592744
- [Background] Senthilvel E, Auckley D, Dasarathy J. Evaluation of sleep disorders in the primary care setting: history taking compared to questionnaires. J Clin Sleep Med. 2011 Feb 15;7(1):41-8. PMID 21344054
- [Background] Auckley D, Ramsammy V, Shalhoub G, Khanna G. Suspected OSA in hospitalized patients: prevalence and potential for adverse events. Sleep 2010; 33:A136
- [Background] Gupta RM, Parvizi J, Hanssen AD, Gay PC. Postoperative complications in patients with obstructive sleep apnea syndrome undergoing hip or knee replacement: a case-control study. Mayo Clin Proc. 2001 Sep;76(9):897-905. doi: 10.4065/76.9.897. PMID 11560300
- [Background] Mooe T, Gullsby S, Rabben T, Eriksson P. Sleep-disordered breathing: a novel predictor of atrial fibrillation after coronary artery bypass surgery. Coron Artery Dis. 1996 Jun;7(6):475-8. PMID 8889364
- [Background] Kaw R, Golish J, Ghamande S, Burgess R, Foldvary N, Walker E. Incremental risk of obstructive sleep apnea on cardiac surgical outcomes. J Cardiovasc Surg (Torino). 2006 Dec;47(6):683-9. PMID 17043616
- [Background] Esclamado RM, Glenn MG, McCulloch TM, Cummings CW. Perioperative complications and risk factors in the surgical treatment of obstructive sleep apnea syndrome. Laryngoscope. 1989 Nov;99(11):1125-9. doi: 10.1288/00005537-198911000-00004. PMID 2530406
- [Background] Catley DM, Thornton C, Jordan C, Lehane JR, Royston D, Jones JG. Pronounced, episodic oxygen desaturation in the postoperative period: its association with ventilatory pattern and analgesic regimen. Anesthesiology. 1985 Jul;63(1):20-8. doi: 10.1097/00000542-198507000-00004. PMID 4014768
- [Background] Sollevi A, Lindahl SG. Hypoxic and hypercapnic ventilatory responses during isoflurane sedation and anaesthesia in women. Acta Anaesthesiol Scand. 1995 Oct;39(7):931-8. doi: 10.1111/j.1399-6576.1995.tb04200.x. PMID 8848894
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. Validation of the Berlin questionnaire and American Society of Anesthesiologists checklist as screening tools for obstructive sleep apnea in surgical patients. Anesthesiology. 2008 May;108(5):822-30. doi: 10.1097/ALN.0b013e31816d91b5. PMID 18431117
- [Background] Flemons WW, Whitelaw WA, Brant R, Remmers JE. Likelihood ratios for a sleep apnea clinical prediction rule. Am J Respir Crit Care Med. 1994 Nov;150(5 Pt 1):1279-85. doi: 10.1164/ajrccm.150.5.7952553.